CLINICAL TRIAL: NCT00336414
Title: Five-Year Single-Blind, Phase III Effectiveness Randomised Actively Controlled Clinical Trial in New Onset Juvenile Systemic Lupus Erythematosus Nephritis: Oral Cyclophosphamide Versus High Dose Intravenous Cyclophosphamide Versus Intermediate Dose Intravenous Cyclophosphamide
Brief Title: Five-Year Actively Controlled Clinical Trial in New Onset Juvenile Systemic Lupus Erythematosus Nephritis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: the study is withdrawn due to low and unexpected enrollment rate
Sponsor: Istituto Giannina Gaslini (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IGG-PRINTO-003
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2007-06

CONDITIONS: Systemic Lupus Erythematosus Nephritis
Keywords: Juvenile Systemic Lupus Erythematosus nephritis; randomised actively controlled clinical trial; cyclophosphamide; prednisone; azathioprine; methylprednisolone

INTERVENTIONS:
Drug: cyclophosphamide-prednisone-azathioprine

SUMMARY:
This is a 5-year project, involving 185 partners from 46 countries (110 in 21 EU States and 75 in 25 extra-EU States), with a randomised clinical trials (RCT) in juvenile systemic lupus erythematosus (JSLE): 5-year phase III single-blind, RCT in children with newly diagnosed, WHO class III, IV JSLE proliferative nephritis: PDN and oral cyclophosphamide (CYC) versus high dose intravenous (iv) CYC versus intermediate dose iv CYC, followed by maintenance with azathioprine.The trial is aimed to find out the treatment regimen associated with the lowest occurrence of flare and the lowest drug related toxicity.

DETAILED DESCRIPTION:
Scientific objectives: The proposed project is aimed to improve treatment approaches for rare, severe and disabling paediatric rheumatic diseases (PRD). This goal will be achieved by the Paediatric Rheumatology International Trials Organisation (PRINTO) an international network whose main function is to provide a scientific base for current PRD treatments for which no evidence based data exist in the literature, and for drugs for which there is no support from industries.

This is a 5-year project, involving 185 partners from 46 countries (110 in 21 EU States and 75 in 25 extra-EU States), with a randomised clinical trials (RCT) in juvenile systemic lupus erythematosus (JSLE): 5-year phase III single-blind, RCT in children with newly diagnosed, WHO class III, IV JSLE proliferative nephritis: PDN and oral cyclophosphamide (CYC) versus high dose intravenous (iv) CYC versus intermediate dose iv CYC, followed by maintenance with azathioprine. The JSLE RCT is aimed to find out the treatment regimen associated with the lowest occurrence of flare and the lowest drug related toxicity. The retention on treatment will be used as main measure of effectiveness.

Methodology: The present protocol is the natural follow up of previous work conducted by PRINTO. In particular the RCT foreseen in this protocol is modelled after the successful completion of an early phase trial with MTX in juvenile idiopathic arthritis, and will use validated JSLE outcome measures for the evaluation of response to therapy.

It is the basic premise of this protocol that, without i) the involvement of the international paediatric rheumatology community, ii) the innovative type of mechanism described herein, these studies would never be conducted.

Objectives. The goals of the current protocol is therefore the natural follow-up of the objectives achieved with the previous grants and, in particular, of projects designed to discern new models for the successful conduct of clinical trials in children with rare diseases, and to develop standardized and validated measures for the evaluation of response to therapy in JSLE.

The proposed trials in in JSLE (oral cyclophosphamide [CYC] versus intermediate dose intravenous [iv] CYC versus high dose iv CYC) followed by maintenance therapy with azathioprine [AZA]), should serve as a model for the successful running of early phase clinical trials for severe and disabling rare diseases of childhood. The ultimate aim of these trials is to provide evidence-based information about the clinical utility of drugs in the management of rare paediatric conditions.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed children with untreated and biopsy proven revised WHO Class III, IV proliferative lupus nephritis and 24 hour proteinuria ≥ 500 mg/day. The kidney biopsy specimen will be read by the renal pathologists of the participating centres (light and immunofluorescence) (54). Slides of paraffin-embedded sections from all patients will be re-viewed by a blinded a renal pathologist at the PRINTO coordinating centre.

Diagnosis of JSLE according to the ACR revised classification criteria (57); Age at enrolment ≤ 18 years. Female of child-bearing potential must have a negative pregnancy test at the beginning of the trial, and then every 3 months. If sexually active, they must agree to use adequate contraception, throughout study participation, and must have no intention of conceiving during the course of the study. Post-pubertal males must have no plans to father a child during the study and agree to use adequate birth control methods if sexually active.

Ability to comply with the entire study procedures, ability to communicate meaningfully with the investigational staff, competence to give written informed consent; to be applied to the parents and/or patients, as appropriate Duly executed, written, informed consent obtained from the parents or other legal representative and/or the patient according to requirement of the local ethics committee.

Exclusion Criteria:

Treatment with the CYC, AZA or mycophenolate mofetil anytime before randomisation.

Neutrophil count <1,500 cell/mm3 and/or platelet count <50,000/mm3. History of poor compliance with previous treatment. Evidence of current use of alcohol or illicit drugs abuse. Live vaccines not allowed during the entire duration of the trial.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Primary: 50% improvement in at least 2 core set variables with no more tha 1 of the remaining variables worsened by> 30%
core set variables:
physician's global assessment of disease activity on a 10 cm visual analogue scale; global disease activity measure by the mean of the European Consensus Lupus Activity parent's/patient's global assessment of overall well-being on a 10 cm VAS;
health-related quality of life assessment.

SECONDARY OUTCOMES:
Change over time in the individual components of the JSLE
core set of variables; time to proteinuria disappearance; frequency of drop-out from
suggested steroids use; frequency of drop-out for inefficacy of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolino Ruperto, MD, MPH, Principal Investigator — Istituto Giannina Gaslini-PRINTO
Locations (1):
- Istituto Giannina Gaslini, Genoa, Italy

REFERENCES:
- [Background] Ruperto N, Ravelli A, Murray KJ, Lovell DJ, Andersson-Gare B, Feldman BM, Garay S, Kuis W, Machado C, Pachman L, Prieur AM, Rider LG, Silverman E, Tsitsami E, Woo P, Giannini EH, Martini A; Paediatric Rheumatology International Trials Organization (PRINTO); Pediatric Rheumatology Collaborative Study Group (PRCSG). Preliminary core sets of measures for disease activity and damage assessment in juvenile systemic lupus erythematosus and juvenile dermatomyositis. Rheumatology (Oxford). 2003 Dec;42(12):1452-9. doi: 10.1093/rheumatology/keg403. Epub 2003 Jun 27. PMID 12832713
- [Background] Ruperto N, Ravelli A, Cuttica R, Espada G, Ozen S, Porras O, Sztajnbok F, Falcini F, Kasapcopur O, Venning H, Bica B, Merino R, Coto C, Ros J, Susic G, Gamir ML, Minden K, See Y, Uziel Y, Mukamel M, Riley P, Zulian F, Olivieri AN, Cimaz R, Girschick H, Rumba I, Cavuto S, Pistorio A, Lovell DJ, Martini A; Pediatric Rheumatology International Trials Organization (PRINTO); Pediatric Rheumatology Collaborative Study Group (PRCSG). The Pediatric Rheumatology International Trials Organization criteria for the evaluation of response to therapy in juvenile systemic lupus erythematosus: prospective validation of the disease activity core set. Arthritis Rheum. 2005 Sep;52(9):2854-64. doi: 10.1002/art.21230. PMID 16142708
- [Background] Ruperto N, Ravelli A, Oliveira S, Alessio M, Mihaylova D, Pasic S, Cortis E, Apaz M, Burgos-Vargas R, Kanakoudi-Tsakalidou F, Norambuena X, Corona F, Gerloni V, Hagelberg S, Aggarwal A, Dolezalova P, Saad CM, Bae SC, Vesely R, Avcin T, Foster H, Duarte C, Herlin T, Horneff G, Lepore L, van Rossum M, Trail L, Pistorio A, Andersson-Gare B, Giannini EH, Martini A; Pediatric Rheumatology International Trials Organization. The Pediatric Rheumatology International Trials Organization/American College of Rheumatology provisional criteria for the evaluation of response to therapy in juvenile systemic lupus erythematosus: prospective validation of the definition of improvement. Arthritis Rheum. 2006 Jun 15;55(3):355-63. doi: 10.1002/art.22002. PMID 16739203
- [Background] Boumpas DT, Austin HA 3rd, Vaughn EM, Klippel JH, Steinberg AD, Yarboro CH, Balow JE. Controlled trial of pulse methylprednisolone versus two regimens of pulse cyclophosphamide in severe lupus nephritis. Lancet. 1992 Sep 26;340(8822):741-5. doi: 10.1016/0140-6736(92)92292-n. PMID 1356175
- [Background] Gourley MF, Austin HA 3rd, Scott D, Yarboro CH, Vaughan EM, Muir J, Boumpas DT, Klippel JH, Balow JE, Steinberg AD. Methylprednisolone and cyclophosphamide, alone or in combination, in patients with lupus nephritis. A randomized, controlled trial. Ann Intern Med. 1996 Oct 1;125(7):549-57. doi: 10.7326/0003-4819-125-7-199610010-00003. PMID 8815753
- [Background] Contreras G, Pardo V, Leclercq B, Lenz O, Tozman E, O'Nan P, Roth D. Sequential therapies for proliferative lupus nephritis. N Engl J Med. 2004 Mar 4;350(10):971-80. doi: 10.1056/NEJMoa031855. PMID 14999109
- [Background] Houssiau FA, Vasconcelos C, D'Cruz D, Sebastiani GD, Garrido Ed Ede R, Danieli MG, Abramovicz D, Blockmans D, Mathieu A, Direskeneli H, Galeazzi M, Gul A, Levy Y, Petera P, Popovic R, Petrovic R, Sinico RA, Cattaneo R, Font J, Depresseux G, Cosyns JP, Cervera R. Immunosuppressive therapy in lupus nephritis: the Euro-Lupus Nephritis Trial, a randomized trial of low-dose versus high-dose intravenous cyclophosphamide. Arthritis Rheum. 2002 Aug;46(8):2121-31. doi: 10.1002/art.10461. PMID 12209517
- [Background] Mok CC, Ho CT, Siu YP, Chan KW, Kwan TH, Lau CS, Wong RW, Au TC. Treatment of diffuse proliferative lupus glomerulonephritis: a comparison of two cyclophosphamide-containing regimens. Am J Kidney Dis. 2001 Aug;38(2):256-64. doi: 10.1053/ajkd.2001.26084. PMID 11479150
- [Background] Yee CS, Gordon C, Dostal C, Petera P, Dadoniene J, Griffiths B, Rozman B, Isenberg DA, Sturfelt G, Nived O, Turney JH, Venalis A, Adu D, Smolen JS, Emery P. EULAR randomised controlled trial of pulse cyclophosphamide and methylprednisolone versus continuous cyclophosphamide and prednisolone followed by azathioprine and prednisolone in lupus nephritis. Ann Rheum Dis. 2004 May;63(5):525-9. doi: 10.1136/ard.2002.003574. PMID 15082482
- See also: Web site of the international network who is conducting the trial — http://www.printo.it